CLINICAL TRIAL: NCT00414726
Title: Clinical Trial of Normobaric Oxygen Therapy in Acute Ischemic Stroke
Brief Title: Normobaric Oxygen Therapy in Acute Ischemic Stroke Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Imbalance in deaths favoring control arm; deaths not attributed to treatment by the blinded external medical monitor.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Aneesh B. Singhal, MD, Associate Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01NS051412 (NIH); P50NS051343 (NIH)
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; normobaric oxygen therapy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NBO (Normobaric Oxygen) (Active Comparator): Oxygen, inhaled at 30-45L/min via a facemask for 8 hours
  Interventions: Drug: NBO (Normobaric Oxygen); Drug: Room Air
- Room Air (Placebo Comparator): Room Air, inhaled at 30-45L/min via a facemask for 8 hours
  Interventions: Drug: NBO (Normobaric Oxygen); Drug: Room Air

INTERVENTIONS:
Drug: NBO (Normobaric Oxygen) — High-flow oxygen delivered via a facemask. A total of 240 individuals with acute ischemic stroke will be randomized 1:1 to receive either room air or oxygen administered at 30-45 L/min via a simple facemask for 8 hours.
Drug: Room Air — Room Air delivered via a facemask. A total of 240 individuals with acute ischemic stroke will be randomized 1:1 to receive either room air or oxygen administered at 30-45 L/min via a simple facemask for 8 hours.

SUMMARY:
The purpose of this study is to compare the safety and efficacy of treating individuals with acute ischemic stroke with normobaric oxygen therapy (NBO, given within 9 hours of symptom onset), to standard medical treatment.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death and the leading cause of disability in the United States. Ischemic stroke is caused by a blockage of blood flow to one or more brain arteries, usually due to a blood clot. As a result there is a reduced supply of oxygen and other nutrients leading to permanent brain damage. Normobaric oxygen therapy (NBO, or high-flow oxygen delivered via a facemask) shows promise as a simple, widely accessible, low-cost therapy that can prevent stroke-related brain damage and extend the time window for administering the clot-busting drug t-PA (tissue plasminogen activator), which is the only acute stroke treatment approved by the Food and Drug Administration.

The primary goal of this trial is to compare the safety and therapeutic efficacy of NBO (started within 9 hours of symptom onset) to standard medical treatment with Room Air. We aim to enroll a total of 240 individuals with acute ischemic stroke less than 9 hours after symptom onset, at the Massachusetts General and Brigham and Women's Hospitals in Boston. Participants will be randomly selected to receive either room air (RA, control) or NBO (active treatment) at flow rates of 30-45L/min administered via a face mask for 8 hours. Neurological function scores and neuroimaging [magnetic resonance imaging (MRI) or computed tomography (CT) scans] will be obtained before, during, and after therapy until 90 days.

This study is part of the Specialized Program of Translational Research in Acute Stroke (SPOTRIAS), which allows researchers to enhance and initiate translational research that ultimately will benefit individuals with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Acute ischemic stroke in whom treatment can potentially be started within 9 hours after symptom onset. If the symptom onset time is unknown, the time of onset will be defined as the midpoint between the time when the subject was last seen neurologically intact, and when found to have a neurological deficit.
* National Institutes of Health Stroke Scale (NIHSS) score 4 or greater.

Exclusion Criteria:

* Patients being actively considered for intravenous or intra-arterial thrombolysis will be excluded.
* Patients likely to have acute stroke intervention such as carotid endarterectomy or stent or angioplasty, hemicraniectomy, etc.
* Rapidly improving neurological deficits (transient ischemic attack).
* Known history of severe chronic obstructive pulmonary disease (Forced Expiratory Vital Capacity less than 1.0 or oxygen dependent).
* More than 3 L/min oxygen required to maintain peripheral arterial oxygen saturation above 92%.
* New York Heart Association Class III heart failure.
* Endotracheal intubation prior to enrollment or impending need for artificial ventilation.
* Coma (National Institutes of Health Stroke Scale item 1a score of 3).
* Suspected seizure at or after onset of stroke, or a known active seizure disorder.
* Blood glucose below 50 mg/dL or greater than 250 mg/dL prior to enrollment.
* Concurrent severe non-stroke medical illness requiring admission to a non-neurological intensive care unit
* Expected survival less than 90 days.
* Any condition that might limit neurological assessment or follow-up in the opinion of the investigator.
* Pre-menopausal women with a positive pregnancy blood test performed at admission.
* Inability to obtain consent from the patient or legally authorized representative.
* Active participation in another intervention study (e.g. investigational drug trial).
* Proven alternate etiology for stroke-like symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aneesh B Singhal, MD, Principal Investigator — Massachusetts General and Brigham & Women's Hospitals
Locations (2):
- United States (2):
  - Massachusetts General Hospital, ACC-729C, Boston, Massachusetts
  - Brigham and Women's Hospital, 75 Francis Street, Boston, Massachusetts

REFERENCES:
- [Background] Singhal AB, Benner T, Roccatagliata L, Koroshetz WJ, Schaefer PW, Lo EH, Buonanno FS, Gonzalez RG, Sorensen AG. A pilot study of normobaric oxygen therapy in acute ischemic stroke. Stroke. 2005 Apr;36(4):797-802. doi: 10.1161/01.STR.0000158914.66827.2e. Epub 2005 Mar 10. PMID 15761201
- [Background] Kim HY, Singhal AB, Lo EH. Normobaric hyperoxia extends the reperfusion window in focal cerebral ischemia. Ann Neurol. 2005 Apr;57(4):571-5. doi: 10.1002/ana.20430. PMID 15786465
- [Background] Singhal AB, Dijkhuizen RM, Rosen BR, Lo EH. Normobaric hyperoxia reduces MRI diffusion abnormalities and infarct size in experimental stroke. Neurology. 2002 Mar 26;58(6):945-52. doi: 10.1212/wnl.58.6.945. PMID 11914413
- [Background] Singhal AB, Ratai E, Benner T, Vangel M, Lee V, Koroshetz WJ, Schaefer PW, Sorensen AG, Gonzalez RG. Magnetic resonance spectroscopy study of oxygen therapy in ischemic stroke. Stroke. 2007 Oct;38(10):2851-4. doi: 10.1161/STROKEAHA.107.487280. Epub 2007 Aug 30. PMID 17761914
- [Background] Singhal AB. Oxygen therapy in stroke: past, present, and future. Int J Stroke. 2006 Nov;1(4):191-200. doi: 10.1111/j.1747-4949.2006.00058.x. PMID 18706016
- [Background] Fujiwara N, Murata Y, Arai K, Egi Y, Lu J, Wu O, Singhal AB, Lo EH. Combination therapy with normobaric oxygen (NBO) plus thrombolysis in experimental ischemic stroke. BMC Neurosci. 2009 Jul 15;10:79. doi: 10.1186/1471-2202-10-79. PMID 19604385
- [Derived] Regenhardt RW, Gonzalez RG, He J, Lev MH, Singhal AB. Symmetric CTA Collaterals Identify Patients with Slow-progressing Stroke Likely to Benefit from Late Thrombectomy. Radiology. 2022 Feb;302(2):400-407. doi: 10.1148/radiol.2021210455. Epub 2021 Nov 2. PMID 34726532
- See also: Specialized Program of Translational Research in Acute Stroke website — http://www.spotrias.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 2007-June 2009
Groups:
- Normobaric Oxygen: Oxygen, inhaled at 30-45L/min via a facemask for 8 hours
Period: Overall Study
Arm/Group | Normobaric Oxygen | Room Air
Started | 43 | 42
Completed | 43 | 41
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normobaric Oxygen | Room Air | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (14) | 73.4 (14) | 73.7 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 17 | 44
  Male | 16 | 25 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 6 | 6
  Not Hispanic or Latino | 42 | 36 | 78
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 40 | 39 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Outcome Measure is a Comparison of the Change in National Institutes of Health Stroke Scale (NIHSS) Scores From Baseline to 24 Hours (After Therapy) in the Two Groups.
Description: The NIHSS score ranges from 0 (best score) to 42 (worst score).
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: 0-24 hour change in NIHSS score
Arm/Group | Normobaric Oxygen | Room Air
Number analyzed (Participants) | 43 | 42
0-24 hour change in NIHSS score | 0.17 [-1.07 to 1.41] | -0.73 [-2.31 to 0.86]
Statistical Analysis 1: Comparison: Normobaric Oxygen vs Room Air; Subjects were analyzed using an intention to treat approach. All subjects were analyzed at 24 hours. For four subjects missing 24-hour NIHSS scores, the change score was given the highest possible value; Test type: Superiority or Other; p = 0.91, Wilcoxon (Mann-Whitney); We used the Van-Elteren extension of the Wilcoxon rank sum test; ajustments made for baseline NIHSS categories (4-11)(12-20)(>20)

2. Primary Outcome: Primary Efficacy Outcome Measure is a Comparison of the Change in National Institutes of Health Stroke Scale (NIHSS) Scores From Baseline to 4 Hours (During Therapy) in the Two Groups.
Description: The NIHSS score ranges from 0 (best score) to 42 (worst score).
Time Frame: 4 hours after starting treatment
Measure: Mean (95% Confidence Interval); unit: 0-4 hour change in NIHSS score
Arm/Group | Normobaric Oxygen | Room Air
Number analyzed (Participants) | 43 | 42
0-4 hour change in NIHSS score | -0.37 [-1.20 to 0.46] | -0.43 [-1.43 to 0.58]
Statistical Analysis 1: Comparison: Normobaric Oxygen vs Room Air; Test type: Superiority or Other; p = 0.68, Wilcoxon (Mann-Whitney); We used the Van Elteren extension of the Wilcoxin rank sum test that adjusts for stratified randomization

ADVERSE EVENTS:
Time Frame: AEs were collected until the final visit at 3 months (range, 75-110 days). All deaths until day 110 were included.
Description: Total 24 deaths: 7 RA, 17 NBO. The blinded external medical monitor did not adjudicte any death as "definitely" or "probably" related to therapy. One death in each arm was adjudicated as "possibly" related to therapy; 6 deaths in the Room Air arm and 16 deaths in the NBO arm, were adjudicated as "unlikely or unrelated" to therapy.
Arm/Group | Normobaric Oxygen | Room Air
Serious Adverse Events (participants affected / at risk) | 24/43 | 20/41
Other Adverse Events (participants affected / at risk) | 42/43 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normobaric Oxygen (N=43) | Room Air (N=41)
Cardiac Arrhythmia (Cardiac disorders) | 1 | 3
Cardiac General (Cardiac disorders) | 3 | 2
Constitutional Symptoms (General disorders) | 0 | 1
Death (General disorders) | 17 | 7
Hemorrhage/Bleeding (General disorders) | 4 | 0
Hepatobiliary/Pancreas (Hepatobiliary disorders) | 1 | 0
Infection (Infections and infestations) | 2 | 1
Metabolic/Laboratory (Investigations) | 0 | 1
Neurology (Nervous system disorders) | 8 | 3
Pain (General disorders) | 1 | 0
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Renal/Genitourinary (Renal and urinary disorders) | 0 | 2
Vascular (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normobaric Oxygen (N=43) | Room Air (N=41)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 5 | 3
Cardiac Arrhythmia (Cardiac disorders) | 9 | 7
Cardiac General (Cardiac disorders) | 12 | 6
Constitutional Symptoms (General disorders) | 16 | 10
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 14 | 11
Gastrointestinal (Gastrointestinal disorders) | 14 | 18
Hemorrhage/Bleeding (General disorders) | 14 | 15
Infection (Infections and infestations) | 16 | 13
Lymphatics (Blood and lymphatic system disorders) | 9 | 7
Metabolic/Laboratory (Investigations) | 4 | 3
Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 0 | 3
Neurology (Nervous system disorders) | 27 | 18
Pain (General disorders) | 18 | 15
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 23 | 13
Renal/Genitourinary (Renal and urinary disorders) | 10 | 11

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No